CLINICAL TRIAL: NCT06725108
Title: Non-invasive Continuous Hemodynamic Monitoring in Acute Brain Injury
Brief Title: Hemodynamic ABI Monitor
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB23-0973
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Brain Injury (TBI); Intracerebral Hemorrhage
Keywords: Hemodynamic; Acute brain injury; Monitoring
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to explore the relationship of heart function with the course and outcomes after traumatic brain injuries and nontraumatic intracerebral hemorrhage. The goal is to explore association between routinely collected hemodynamic and brain monitoring data.

Participants already taking intervention A as part of their regular medical care and the investigators will follow up with participants 6 months after discharging the hospital.

DETAILED DESCRIPTION:
This is a prospective observational study collecting data produced as part of standard routine clinical care and the study team will collect the data from Starling Monitor and subject medical record. Adult patients undergoing hemodynamic monitoring with the Starling monitor as part of their standard of care will be considered as a candidate for the study. Patients will only be included in this study if they agree to take part in the data collection. If the patient declines participation, they will still undergo hemodynamic monitoring with the Starling hemodynamic monitor, but their clinical and Starling device information will not be collected to be entered into the database.

No clinical interventions are part of the study. There is no interference of data collected with clinical decision making. Hemodynamic data will be derived via the application of the entirely non-invasive, FDA approved for clinical use, Starling System (provided by Baxter for this study).

Prior to enrollment, the study team will provide patients and/or their family members the details of the study, answer any questions and address concerns. The patient and/or their families will then be given time to consider participation. After informed consent is obtained from the patient or legally authorized representative, patient data will be extracted from the electronic medical record (EMR) into a REDCap database and Case Report Forms (CRFs).

The study team also will collect the data from the Starling Monitor and subject's medical record.

Data collection:

Case Report Forms (CRFs) will be used to collect all patient data during the course of the study and will be entered into an electronic database. Data will be collected on patients from the initiation to completion of monitoring with the Starling Monitor. The occurrence of any advice related Adverse Events will be collected throughout this period.

The following data will be collected by chart review:

* demographics
* risk factors
* diagnoses
* medical surgical treatments
* laboratory imaging studies
* Changes in hemodynamics
* treatment and outcome for patients with TBI
* Volume of fluid administered
* Percent of patients that are fluid responsive
* Incidence of diastolic dysfunction
* % fluid responsiveness in diastolic dysfunction
* Days on ventilator
* Days on vasopressors
* cerebral hemodynamics: intracranial pressure (ICP), cerebral perfusion pressure (CPP), partial brain tissue oxygenation (PbtO2), and cerebral blood flow (CBF)

The following data will be summarized descriptively:

* Treatment details (intervention, intubation, ventilation, start of a new medication)
* Medications
* Volume of fluid administered
* Demographics, such as patient diagnosis
* Setting
* Fluid bolus assessment, if applicable
* Additional hemodynamic assessment methods, if utilized
* Patient outcome data
* cerebral hemodynamics: intracranial pressure (ICP), cerebral perfusion pressure (CPP), partial brain tissue oxygenation (PbtO2), and CBF

Follow-up medical history will be obtained at 180 days via the EMR or patient report. Primary endpoints are functional outcomes and quality of life at 180 days after hospital discharge. The follow-up functional status and quality of life measures will be done by telephone, in-person at their regularly scheduled follow-up appointment, or by email, for less than 30 minutes using validated instruments and/or using a web-based REDCap survey. However, these surveys can also be completed during the subject's 180-day follow up visit with their doctor or a telephone follow-up. The follow up telephone call/visit will last for less than 30 minutes and will consist of a series of validated instruments/questionnaires. The following instruments will be used:

Glasgow Outcome Scale Extended (GOSE) to ascertain functional status

The goal is to examine the association between systemic hemodynamics, cerebral hemodynamics, clinical management parameters, and clinical outcomes in patients with severe traumatic brain injury and nontraumatic intracerebral hemorrhage. Specifically, we are interested in Cardiac index, fluid responsiveness (FR) markers, fluid balance, hemodynamic support, and intensive care unit (ICU) mortality and functional outcome at 6 months, measured by the Glasgow Outcome Scale Extended (GOSE). Patient-level analyses will involve adjusting for key characteristics per patient, such as IMPACT score, post-resuscitation Glasgow Coma Scale (GCS), and Rotterdam CT classification. For patient-level analyses, random-effects logistic regression (for ICU mortality) and ordinal regression (for GOSE) will be used, with adjustment for IMPACT variables, major extracranial injuries, and Rotterdam Computed Tomography (CT) scale. Additionally, the study will explore the relationships between systemic and cerebral hemodynamics. Continuous variables will be reported as median with interquartile range (IQR), while binomial variables will be presented as counts with percentages (%). Statistical tests, such as the Wilcoxon-Mann Whitney test for continuous variables and Fisher's-exact test for categorical variables, will be performed to compare the groups. To assess the association of identified variables with neurologic outcomes, univariate logistic regression models will be used. Subsequently, a multivariate logistic regression model will be employed to determine the independent variables associated with mortality and neurologic outcomes.

To explore the temporal relationships and directions of change among systemic and cerebral hemodynamic time series data, Granger causality testing will be applied.

ELIGIBILITY:
Inclusion:

Patients who are:

* Admitted to the University of Chicago Medical Center Neurocritical Care Unit
* Adults between 18 years and 80
* Admitted with Traumatic brain injury blunt and penetrating or nontraumatic intracerebral hemorrhage
* post-resuscitation Glasgow Coma Scale (GCS) <9

Exclusion:

Patients who were:

* Pre-existing heart failure
* Moribund or neurological exam suggesting imminent brain death (bilateral, fixed and dilated pupils) on admission
* Major polytrauma or admitted to the surgical trauma critical care service
* Prisoner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to the University of Chicago Medical Center Neurocritical Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
functional outcomes | 180 days after discharging the hospital
  Primary endpoints are functional outcomes and quality of life at 180 days after hospital discharge. The follow-up functional status and quality of life measures will be done by telephone, in-person at their regularly scheduled follow-up appointment, or by email, for less than 30 minutes using validated instruments and/or using a web-based REDCap survey. However, these surveys can also be completed during the subject's 180-day follow up visit with their doctor or a telephone follow-up. The follow up telephone call/visit will last for less than 30 minutes and will consist of a series of validated instruments/questionnaires. The following instruments will be used:
  Glasgow Outcome Scale Extended (GOSE) to ascertain functional status The GOSE score ranges from 1 to 8, with the minimum score of 1 indicating Death and the highest score of 8 representing a Good Recovery, signifying a good outcome and a return to pre-injury functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Lazaridis, MD, Principal Investigator — university of Chicago attending
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided